CLINICAL TRIAL: NCT06491667
Title: Neutrophil-to-Lymphocyte Ratio AND C-REATIVE PROTEIN Useful as Cost-Effective Preliminary Prognostic Markers in ST-Elevation Myocardial Infarction
Brief Title: NLR AND CRP Useful as Cost-Effective Preliminary Prognostic Markers in ST-Elevation Myocardial Infarction
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Albier Youssef Kaiser, Resident at Internal Medicine Department Sohag University hospital, Sohag University
Other Study IDs: Soh-med-24-0614MS
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Elevated NLR and CRP level: Elevated NLR and CRP level
  Interventions: Diagnostic Test: CBC; Diagnostic Test: C-reactive protein
- Normal NLR and CRP level: Elevated NLR and CRP level
  Interventions: Diagnostic Test: CBC; Diagnostic Test: C-reactive protein

INTERVENTIONS:
Diagnostic Test: CBC — Explore the role of Neutrophil-lymphocyte ratio C-reactive protein in predicting the imediate and short-term prognosis in ST-segment elevation myocardial infarction
Diagnostic Test: C-reactive protein — Explore the role of Neutrophil-lymphocyte ratio C-reactive protein in predicting the imediate and short-term prognosis in ST-segment elevation myocardial infarction

SUMMARY:
Acute myocardial infarction (AMI) is a serious and fatal cardiovascular emergency and considered the leading cause of mortality worldwide.

Atherosclerosis of coronary arteries which takes decades to manifest clinically, is the primary predisposing pathologic factor responsible for the development of coronary heart disease It has been shown that A complex immune and inflammatory pathophysiological process is thought to be crucial for in the initiation and progression of atherosclerotic plaques.

Inflammation is one of the main mechanisms in the pathogenesis of atherosclerosis , Destabilization of chronic artery plaques and development of thrombosis, which are the main mechanisms in the pathophysiology of ST-segment elevation myocardial infarction (STEMI).

, and the interest to the evaluation of inflammatory biomarkers in coronary artery disease (CAD) has been increasing over the last decade .

Although numerous inflammatory markers, including troponin T/I, lactate dehydrogenase (LDH), and creatine kinase (CK-MB), are linked to worsened clinical outcomes in both ST elevation and non-ST elevation myocardial infarction (NSTEMI), there is an unmet need for a cost-effective biomarker for impoverished countries of the world .

The neutrophil-to-lymphocyte ratio (NLR), and C-reactive protein (CRP) ; has emerged as an important inflammatory markers for cardiovascular risk stratification.

And are relatively cheap inflammatory markers, can act as a bridge to mitigate the gap in assessing the cardiovascular risk and outcomes

DETAILED DESCRIPTION:
Acute myocardial infarction (AMI) is a serious and fatal cardiovascular emergency and considered the leading cause of mortality worldwide.

* Atherosclerosis of coronary arteries which takes decades to manifest clinically, is the primary predisposing pathologic factor responsible for the development of coronary heart disease
* It has been shown that A complex immune and inflammatory pathophysiological process is thought to be crucial for in the initiation and progression of atherosclerotic plaques
* Inflammation is one of the main mechanisms in the pathogenesis of atherosclerosis , Destabilization of chronic artery plaques and development of thrombosis, which are the main mechanisms in the pathophysiology of ST-segment elevation myocardial infarction (STEMI) .

  , and the interest to the evaluation of inflammatory biomarkers in coronary artery disease (CAD) has been increasing over the last decade .
* Although numerous inflammatory markers, including troponin T/I, lactate dehydrogenase (LDH), and creatine kinase (CK-MB), are linked to worsened clinical outcomes in both ST elevation and non-ST elevation myocardial infarction (NSTEMI), there is an unmet need for a cost-effective biomarker for impoverished countries of the world
* The neutrophil-to-lymphocyte ratio (NLR), and C-reactive protein (CRP) ;
* has emerged as an important inflammatory markers for cardiovascular risk stratification.
* And are relatively cheap inflammatory markers, can act as a bridge to mitigate the gap in assessing the cardiovascular risk and outcomes In patients with acute myocardial infarction.
* Recent data indicates a strong independent relationship between increased complications after acute myocardial infarction in patients with a high NLR and high CRP level at admission and the initial post-hospitalization period.
* Accordingly, we designed this study to assess the predictive value and prognosis of NLR and CRP in ST-elevation myocardial infarction (STEMI).

ELIGIBILITY:
Inclusion Criteria:

* Patients with age ≥18 years of either sex, with either increase in serum cardiac biomarkers or ECG are STEMI.

Exclusion Criteria:

* Patients presenting with NSTEMI and unstable angina
* Patients with any of these associated conditions that can affect NLR or CRP including
* Inflammatory conditions such as collagen-vascular disorders
* Acute or chronic infectious diseases.
* Auto-immune and neoplastic diseases.
* Chronic hepatic diseases.
* Renal failure.
* Thyroid disorders.
* Previous valvular heart disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: - Patients with age ≥18 years of either sex, with either increase in serum cardiac biomarkers or ECG are STEMI
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Neutrophil-lymphocyte ratio | 6 months
  Explore the role of Neutrophil-lymphocyte ratio in predicting the imediate and short-term prognosis in ST-segment elevation myocardial infarction
C-reactive protein | 6 months
  C-reactive protein in predicting the imediate and short-term prognosis in ST-segment elevation myocardial infarction

CONTACTS AND LOCATIONS:
Overall Officials: Magdy M Amin, Professor, Principal Investigator — Sohag University
Locations (1):
- Sohag university hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Gualandro DM, Caramelli B, Yu PC, Marques AC, Calderaro D. Perioperative myocardial infarction has been forgotten. J Am Coll Cardiol. 2008 May 6;51(18):1825-6; author reply 1826. doi: 10.1016/j.jacc.2008.01.035. No abstract available. PMID 18452792
- [Result] Sahoo S, Losordo DW. Exosomes and cardiac repair after myocardial infarction. Circ Res. 2014 Jan 17;114(2):333-44. doi: 10.1161/CIRCRESAHA.114.300639. PMID 24436429
- [Result] Kuklina EV, Yoon PW, Keenan NL. Prevalence of coronary heart disease risk factors and screening for high cholesterol levels among young adults, United States, 1999-2006. Ann Fam Med. 2010 Jul-Aug;8(4):327-33. doi: 10.1370/afm.1137. PMID 20644187
- [Result] Libby P, Ridker PM, Maseri A. Inflammation and atherosclerosis. Circulation. 2002 Mar 5;105(9):1135-43. doi: 10.1161/hc0902.104353. PMID 11877368